CLINICAL TRIAL: NCT04926662
Title: Understanding Rural Patient and Provide Preferences for Mobile Lung Cancer Screening Clinics
Status: Suspended | Type: Observational
Why Stopped: Study is paused while pre-aim 1 work is being done
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, David J. Finley, Staff Physician, Thoracic Surgery, Dartmouth-Hitchcock Medical Center
Other Study IDs: D21031
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Aim 1: Focus Groups: Focus groups will be conducted in 2 New Hampshire and 2 Vermont towns to better understand patient knowledge, attitudes, and preferences regarding access to lung cancer screening.
- Aim 2: Cross Sectional Survey: Based on focus group feedback, the investigators will visit each proposed site to survey on 2 separate dates to confirm days and times of high traffic. The investigators will also survey patrons at the proposed locations to further determine prospective patient mobile screening preferences and evaluate willingness to participate in screening.
- Aim 3: Survey with follow up data: The investigators will pilot mobile lung cancer screening clinics at each chosen location using the knowledge acquired from focus group experience and local patient survey. Surveys will be conducted at these clinics, and patients will be followed for up to 5 years.

SUMMARY:
The purpose of this study is to research patient preferences for lung cancer screening and pilot mobile units to address the barrier of access that decreases participation in lung cancer screening.

DETAILED DESCRIPTION:
The overarching goal of this study is to research patient preferences for lung cancer screening and pilot mobile units to address the barrier of access that decreases participation in lung cancer screening. To facilitate this, the investigators will evaluate the feasibility of mobile lung cancer screening clinics to improve access through focus group study in designated rural areas of New Hampshire and Vermont, canvas and survey these areas to confirm need, and pilot the mobile lung cancer screening clinic to establish practicability. Findings from the proposed project will be used as preliminary data to apply for further funding and to implement the mobile unit in these identified rural communities on a consistent basis.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 50 to 80 years old
* 20 pack-year smoking history who are currently smoking or have quit smoking within the last 15 years

Exclusion Criteria:

-

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The individuals that will be included in this study will be those that meet lung cancer screening eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 6 months after starting the mobile lung cancer screening units (Aim 3)
  Number of individuals recruited to the mobile lung cancer screening units

SECONDARY OUTCOMES:
Change in knowledge | 6 months after starting the mobile lung cancer screening units (Aim 3)
  Change in knowledge before and after entering the mobile lung cancer screening, as determined by the pre and post survey

CONTACTS AND LOCATIONS:
Overall Officials: David Finley, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Odahowski CL, Zahnd WE, Eberth JM. Challenges and Opportunities for Lung Cancer Screening in Rural America. J Am Coll Radiol. 2019 Apr;16(4 Pt B):590-595. doi: 10.1016/j.jacr.2019.01.001. PMID 30947892
- [Background] Brenner AT, Malo TL, Margolis M, Elston Lafata J, James S, Vu MB, Reuland DS. Evaluating Shared Decision Making for Lung Cancer Screening. JAMA Intern Med. 2018 Oct 1;178(10):1311-1316. doi: 10.1001/jamainternmed.2018.3054. PMID 30105393
- [Background] Atkins GT, Kim T, Munson J. Residence in Rural Areas of the United States and Lung Cancer Mortality. Disease Incidence, Treatment Disparities, and Stage-Specific Survival. Ann Am Thorac Soc. 2017 Mar;14(3):403-411. doi: 10.1513/AnnalsATS.201606-469OC. PMID 28118039
- [Background] Greenwald ZR, El-Zein M, Bouten S, Ensha H, Vazquez FL, Franco EL. Mobile Screening Units for the Early Detection of Cancer: A Systematic Review. Cancer Epidemiol Biomarkers Prev. 2017 Dec;26(12):1679-1694. doi: 10.1158/1055-9965.EPI-17-0454. Epub 2017 Oct 4. PMID 28978564
- [Background] Bhatt S, Isaac R, Finkel M, Evans J, Grant L, Paul B, Weller D. Mobile technology and cancer screening: Lessons from rural India. J Glob Health. 2018 Dec;8(2):020421. doi: 10.7189/jogh.08.020421. PMID 30603075
- [Background] Vang S, Margolies LR, Jandorf L. Mobile Mammography Participation Among Medically Underserved Women: A Systematic Review. Prev Chronic Dis. 2018 Nov 15;15:E140. doi: 10.5888/pcd15.180291. PMID 30447104